CLINICAL TRIAL: NCT06505421
Title: The Effect of Lower Extremity Eccentric Resistance Training on Fatigue in Multiple Sclerosis
Brief Title: Eccentric Exercise and Fatigue in Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Herb Karpatkin, Associate professor, City University of New York, School of Public Health
Other Study IDs: 20240244
Record Dates: First submitted 2024-07-03; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: Exercise; resistance training
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with Multiple sclerosis: Eccentric resistance training , traditional resistance training
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — Eccentric resistance training and tradional resistance training

SUMMARY:
The goal of this observational study is to compare the impact of eccentric resistance training to traditional resistance training on fatigue in persons with multiple sclerosis (MS). The primary question this study is asking is the following: is eccentric resistance training more fatiguing than traditional resistance training in persons with MS?. Participants will be asked to come for two sessions for two weeks. In the first week, subjects will undergo a bout of either traditional or eccentric resistance training. The next day they will return to assess their level of fatigue. The following week the subject will return and undergo whatever type of training they did not experience the first week, and it's effects on fatigue will again be assessed. The difference between the subjects level of fatigue for either condition will be compared.

DETAILED DESCRIPTION:
Persons with multiple sclerosis (MS) have mobility deficits. Exercise is commonly used to treat these mobility deficits, but must be done so judiciously in order to limit the effects of fatigue, one of the most common disease findings. In persons with MS ,fatigue can limit the amount of exercise performed. Eccentric training, where a muscle is lengthened under resistance has been shown to produce greater gains in strength with less energy expenditure when compared to traditional strength training where a muscle is both lengthened and shortened under resistance. However, eccentric strength training has been shown to result in delayed onset muscle soreness, which may also limit how much exercise a person with MS can perform. The purpose of the study is to compare the impact of eccentric versus traditional strength training programs on fatigue and persons with multiple sclerosis. The hypothesis is that there will be no difference in fatigue measurements between the two conditions. If the hypothesis is correct, it will suggest that eccentric training should be the subject of further study to assess it's feasibility and effectiveness, in treating mobility deficits in person with multiple sclerosis.

A randomized crossover design will be used. Ambulatory participants with a diagnosis of MS will be randomized into either a eccentric or traditional training condition. Each training condition will consist of a single session of training. The following day, the patient will return and their levels of fatigue assessed. The next week, the subjects will return and crossover, undergoing whatever type of training they did not experience in the previous week, and the impact of the training will again be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of Multiple Sclerosis.
* Ability to walk for 6 minutes continuously with or without assistive device
* Ability read, understand and sign and informed consent

Exclusion Criteria:

* Evidence of recent exacerbation in the last 2 months prior to starting the study
* Orthopedic, cardiopulmonary, or non -MS neurologic condition that could interfere with carrying out the study protocol

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ambulatory persons with MS
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
6-Minute walk test | Pre-intervention and post intervention for each condition (eccentric and traditional strength training). There is a 36-48 hour period between the pre-intervention and post intervention for each condition
  Subject walks at best possible pace with or without assistive device for 6 minutes. Total distance walked as well as distance per minute is measured

SECONDARY OUTCOMES:
Visual analog scale of fatigue | Pre-intervention and post-intervention for each condition (eccentric vs traditional strength training). There is a 36-48 hour period between the pre-intervention and post intervention for each condition
  Immediately before and after each 6 minute walk subjects will make a mark on a 100mm line indicating their level of fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter College, Physical Therapy Department, City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patrocinio de Oliveira CE, Moreira OC, Carrion-Yagual ZM, Medina-Perez C, de Paz JA. Effects of Classic Progressive Resistance Training Versus Eccentric-Enhanced Resistance Training in People With Multiple Sclerosis. Arch Phys Med Rehabil. 2018 May;99(5):819-825. doi: 10.1016/j.apmr.2017.10.021. Epub 2017 Nov 27. PMID 29191417
- [Background] Wochatz M, Schraplau A, Engel T, Zecher MM, Sharon H, Alt Y, Mayer F, Kalron A. Application of eccentric training in various clinical populations: Protocol for a multi-centered pilot and feasibility study in people with low back pain and people with multiple sclerosis. PLoS One. 2022 Dec 22;17(12):e0270875. doi: 10.1371/journal.pone.0270875. eCollection 2022. PMID 36548298
- [Background] Gauche E, Couturier A, Lepers R, Michaut A, Rabita G, Hausswirth C. Neuromuscular fatigue following high versus low-intensity eccentric exercise of biceps brachii muscle. J Electromyogr Kinesiol. 2009 Dec;19(6):e481-6. doi: 10.1016/j.jelekin.2009.01.006. Epub 2009 Feb 12. PMID 19217311